CLINICAL TRIAL: NCT04730583
Title: Tolerability of Device Based Therapies for Neurofibromatosis Type 1 Cutaneous Neurofibromas
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Massachusetts General Hospital (Other)
Collaborators: Johns Hopkins University (Other)
Responsible Party: Principal Investigator, Richard Rox Anderson, MD, Principle Investigator, Massachusetts General Hospital
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Other
Other Study IDs: 2020P004137
Record Dates: First submitted 2021-01-12; First posted 2021-01-29 (Actual); Last update posted 2025-02-21 (Actual); Status verified 2025-02

CONDITIONS: Cutaneous Neurofibroma
Keywords: Neurofibromatosis Type 1
MeSH Terms: conditions — Neurofibromatosis 1 | interventions — Deoxycholic Acid; Lasers; Lasers, Solid-State

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: Yes | US Export: Yes

ARMS (3):
- Kybella Injection (Active Comparator)
  Interventions: Drug: Kybella
- 1064nm laser (Active Comparator)
  Interventions: Device: 1064nm laser
- 755nm laser (Active Comparator)
  Interventions: Device: 755nm Alexandrite Laser

INTERVENTIONS:
Drug: Kybella — Injection into the cutaneous Neurofibromas lesion
  Arms: Kybella Injection
Device: 1064nm laser — Pulse laser at a wavelength of 1064nm to the cutaneous Neurofibromas lesion
  Arms: 1064nm laser
Device: 755nm Alexandrite Laser — Pulse laser at a wavelength of 755nm to the cutaneous Neurofibromas lesion
  Arms: 755nm laser

SUMMARY:
This study will evaluate the tolerability and effectiveness of three FDA-approved treatments in Neurofibromatosis Type 1 Cutaneous Neurofibromas. These treatments are: a 1064nm laser, a 755nm laser, and a Kybella injection. Each patient will have a treatment and a control site.

ELIGIBILITY:
Inclusion Criteria:

* Adult males and females ≥18 years of age
* Have a diagnosis of Neurofibromatosis Type 1
* Patients must be seeking treatment for cutaneous Neurofibromas
* Patients must have ≥ 6 paired cutaneous Neurofibromas (3 to be treated and 3 untreated) that are visible and measure between 2-4mm in size.
* Able and willing to comply with all visit, treatment and evaluation schedules and requirements
* Able to understand and provide written informed consent
* Access to a Smart Phone to be able to take and upload photographs to an application

Exclusion Criteria:

* Patients who are undergoing other treatment modalities or investigational agents for their cNF lesions
* Individuals who cannot give informed consent or adhere to study schedule
* Actively tanning during the course of the study
* Adverse reactions to compounds of any external agent (e.g., gels, lotions or anesthetic creams) required for use in the study, if no alternative to the said agent exists;
* Known allergy to injectable anesthetics or deoxycholic acid
* Any condition which, in the Investigator's opinion, would make it unsafe (for the participant or study personnel) to treat the participant as part of this research study;
* Pregnant females, due to possible discomfort with the procedure even though the procedure is localized and there is no new drug.

Ages: 18 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 34 (Actual)
Dates: Start 2021-06-02 (Actual); Primary Completion 2024-04-19 (Actual); Study Completion 2024-04-19 (Actual)

PRIMARY OUTCOMES:
Incidence of Treatment-Emergent Adverse Events [Safety and Tolerability] | 3 months after treatment
  Device based treatment will be considered tolerable if <40% of participants treated have a >grade 2 adverse event (AE). A grade 2 AE is defined as an event that requires treatment.

SECONDARY OUTCOMES:
Patient Report Outcomes | For the 12 months after treatment
  Using questionnaires we will determine the patients reported outcomes
Clinician Reported Outcomes | For the 12 months after treatment
  Using questionnaires we will determine the clinicians reported outcomes

CONTACTS AND LOCATIONS:
Overall Officials: R. Rox Anderson, MD, Principal Investigator — Wellman Center for Photomedicine, Massachusetts General Hospital
Locations (1):
- Wellman Center for Photomedicine, Massachusetts General Hospital, Boston, Massachusetts, United States

IPD SHARING:
Plan to Share IPD: No